CLINICAL TRIAL: NCT00420836
Title: Crossover Pharmacokinetic Study of Tobramycin Administered for Inhalation by PARI eFlow® Rapid Electronic Nebulizer (no Compressor) vs. PARI LC PLUSTM Jet Nebulizer (With Compressor) in Cystic Fibrosis Subjects
Brief Title: Tobramycin Administered by eFlow Rapid Nebulizer: Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTBM100B2201
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis, tobramycin, PARI eFlow, PARI LC Plus, nebulizer, pharmacokinetic
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tobramycin

INTERVENTIONS:
Drug: Tobramycin

SUMMARY:
This study assesses the aerosol delivery characteristics (measured by nebulization time, serum and sputum tobramycin pharmacokinetic parameters) and safety of tobramycin administered for inhalation by PARI eFlow rapid electronic nebulizer (no compressor) vs. PARI LC PLUS Jet Nebulizer (with compressor) in subjects with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 6 years or over at the time of screening,
* Chronically colonized with Pseudomonas aeruginosa.
* Diagnosis of cystic fibrosis (CF)
* Ability to expectorate sputum samples on command.
* Ability to tolerate a 1-week washout interval with no inhaled tobramycin or other aminoglycoside treatment.
* Clinically stable in the opinion of the investigator.

Exclusion Criteria:

* Inhaled or intravenous aminoglycosides within 7 days before study drug administration.
* Any investigational drug within 2 weeks before screening.
* Loop diuretics within 7 days before study drug administration.
* Current use of inhaled tobramycin delivered by the PARI LC PLUS jet nebulizer without washout period of at least 1 week before entering the study.
* Women who are, or plan to become, pregnant during the course of the study.
* Serum creatinine or blood urea (BU) above the upper limit of normal for sex and age, or an abnormal urine analysis
* Known local or systemic hypersensitivity to aminoglycosides.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2006-04

PRIMARY OUTCOMES:
Aerosol delivery characteristics of tobramycin when inhaled using either PARI LC PLUS jet nebulizer or PARI eFlow rapid Electronic Nebulizer evaluated by serum concentrations

SECONDARY OUTCOMES:
Potential accumulation of tobramycin in serum measured as the change in tobramycin levels from the first day of treatment to the last day of treatment.
Pharmacokinetics
Safety assessed by adverse events, serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Basel, Study Director — Novartis Pharmaceuticals